CLINICAL TRIAL: NCT06849414
Title: The Relationship Between Blood Homocysteine Level and Motor and Cognitive Manifestation of Parkinson's Disease Patients
Brief Title: The Relationship Between Homocysteine and Manifestation of Parkinson's Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shrouk Mohammed Hossam Eldien Abdelmohsen, principle investigator, Assiut University
Other Study IDs: Homocysteine in PD
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1-First group will include the control group (22) 2- Second group will include PD patients: 22 people will be included in the control group who don't have PD and 22 patients with PD will be enrolled from the clinic of movement disorders of neuropsychiatry hospital of Assiut University and divided into early PD less than 3 years and late more than 3 years
- 1-First group will include the control group (22): 2-Second will include PD patients (22) whose will be collected from the clinic of movement disorders of Neuropsychiatry hospital of Assiut University and then divided into :a-early PD less than 3 years b-late PD more than 3 years

SUMMARY:
* The aim of the current study is to investigate the association between blood homocysteine level and motor as well as cognitive manifestation of PD patients in Assiut governorate.
* Secondary goal is to investigate the association between levels of serum ferritin, iron as well as acute phase proteins (fibrinogen, D-dimer, CRP) and manifestation of PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common progressive neurodegenerative disease which severely affect the quality of life.It was first described by James Parkinson in 1817 as the most prevalent movement disorder and the second most common neurodegenerative disease after Alzheimer's disease (AD).

The etiology of PD remains largely elusive, and the majority of PD cases are of unknown cause.

Homocysteine is included in the pathogenesis of neurodegenerative diseases including PD. Also, patients with hyperhomocysteinemia are more prone to depression and cognitive impairment .Homocysteine is implicated in neurodegenerative diseases via inflammatory response and oxidative stress.

Several studies indicated that iron metabolism is dysregulated in PD. An important fact is the iron loading in dopaminergic neurons of the substantia nigra pars compacta (SNc), which are the cells primarily affected in PD leading to increased neuronal iron and iron-mediated reactive oxygen species (ROS) generation .

Increased Hcy level can facilitate pathological aggregation of proteins involved in neurodegenerative disorders and be toxic to dopaminergic neurons as α synuclein. Homocysteine can modify α synuclein to form more toxic fibrils that are resistant to digestion by proteinases and exhibit propagation activity.

D-dimer serve as risk factor for development of deep venous thrombosis (DVT) in patients with early PD.

Fibrinogen play a role in exacerbating the neuropathological features of neurodegenerative diseases such as PD through regulating pathophysiological mechanisms and signaling pathways while depletion of fibrinogen helps to ameliorate cognitive function impairment in those patients.

ELIGIBILITY:
Inclusion Criteria:

* 1-Inpatients or outpatients from the clinic of movement disorders of neuropsychiatry hospital of Assiut university 2-The age group of the patients is those above 40 years

Exclusion Criteria:

* 1-Secondary parkinsonism associated with specific causes such as infections, medication-induced, poisoning, cerebral arteriosclerosis, and trauma 2-Parkinsonism accompanied by other neurodegenerative disease ( specifically multiple syste atrophy, progressive supranuclear palsy, and dementia with Lewy bodies).

  3-Presence of significant memory or cognitive decline preceding the onset of PD symptoms, as reported by both the patient and/or family members 4-Significant intracranial lesions detected on brain MRI 5-Unable to cooperate in completing the clinical scale assessment and blood sample collection.

  6-Recent or current use of medications such as antiepileptic drugs and certain chemotherapy drugs that can impact blood Hcy levels or the presence of thyroid dysfunction or renal insufficiency that affects Hcy metabolism.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 44 population divided into 22 control and 22 PD patients Informed written consent will be obtained from all participants after explaining the aim of the study to them, and the study will be approved by the ethical committee of our institution
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To investigate the relationship between homocysteine level and motor as well as cognitive manifestation of Parkinson's disease patients | one year